CLINICAL TRIAL: NCT04788966
Title: Evaluation of an Innovative Speech-enabled Translator in Emergency Settings
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Antony Janakiram, Research Assistant, University Hospital, Geneva
Other Study IDs: Réq 2017-00996
Record Dates: First submitted 2021-02-19; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Diagnoses Disease
Keywords: Translation tool; Anamnesis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: the translation tool BabelDr — Doctors use a speech-enabled fixed-phrase translation tool to help communicate with an allophone patient.

SUMMARY:
Survey-based satisfaction, performance and technical features evaluation of a speech-enabled fixed-phrase translation tool (BabelDR) in an emergency department.

ELIGIBILITY:
Inclusion Criteria:

* As per inclusion criteria, patients were required to have no understanding of French, thus making a diagnostic interview by the doctors impossible.

Exclusion Criteria:

* Exclusion criteria concerned patients who shared a common language with the doctor and/or were not able to read in their native language.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients were recruited with an average age of M=38.2 (SD=16.49) of which 53.33% were males. The distribution between the different languages was the following: Spanish (11), Arabic (4), Farsi (7), Tigrinya (7) and Albanian (1).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Satisfaction evaluation through a 4-point scale survey | During the consultation
  Are patients' and doctors' satisfied with the use of BabelDr?
Efficacy evaluation through a 2-point scale survey | During the consultation
  Can BabelDr be efficient tool in an emergency context: are doctors' able to reach a diagnostic with the tool?
Technical features evaluation through a 4-point scale survey | During the consultation
  Are the technical features appreciated by the doctors'?

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided